CLINICAL TRIAL: NCT04863781
Title: Reducing Health Disparities Among African American Women: a Mobile Cognitive Behavioral Stress Management Intervention
Brief Title: Mobile Stress Management Program for African American Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: ISA Associates, Inc. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MD014077
Record Dates: First submitted 2021-04-22; First posted 2021-04-28 (Actual); Last update posted 2024-10-01 (Actual); Status verified 2023-04

CONDITIONS: Psychological Stress
MeSH Terms: conditions — Stress, Psychological

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention (Experimental): All 11 modules will include the following elements: introduction to the topic; two types of assessments (1) adherence to at-home relaxation training practice (following week 2) and (2) 3-5 topic-specific questions to tailor video-based content; a cognitive component; a relaxation component; and a wrap up that includes a brief assessment of module comprehension. Each user will view 5-7 videos per module. Videos will be tailored to user and will last between 2 and 4 minutes. Total time per module will be 20 to 30 minutes. Between modules, users will receive (based on their timing preferences) supportive texts intended to motivate continued engagement or to affirm the life experiences of African American women
  Interventions: Behavioral: Mobile cognitive-behavioral stress management intervention
- Control (Active Comparator): Two mobile courses: Introduction to Stress Management and Techniques for Coping with Stress. Users will be informed that the courses will be completed on their phone, that they are video-based, and that they should spend between 20 and 30 minutes each week, for the next 11 weeks, learning the material. The introductory course defines stress, describes the different sources of stress, and the influence of personality on stress. The coping module includes training in cognitive coping skills, guided imagery, progressive relaxation, autogenic training, and the importance of physical activity to manage stress. All lessons include course assessments. During the intervention period, controls will receive weekly text messages encouraging completion of material.
  Interventions: Behavioral: Control

INTERVENTIONS:
Behavioral: Mobile cognitive-behavioral stress management intervention — Each weekly module will consist of a cognitive component and a relaxation component. The cognitive component during the first 3 weeks will educate users about the Transactional Model of Stress, that discrimination is a type of stressor, and the impact of stress on health. Building on this information, users will then learn how to match coping responses to the changeability of stressors during weeks 4 and 5. The cognitive component will conclude by focusing on the four most common coping strategies used by African American women in response to stress. Modules 2 through 4 will teach progressive muscle relaxation through a series of tension and relaxation cycles. Modules 5 through 8 will train users in diaphragmatic breathing. Finally, users will be trained in three types of mindfulness mediations.
  Arms: Intervention
Behavioral: Control — The introductory course defines stress, describes the different sources of stress, and the influence of personality on stress. The coping module includes training in cognitive coping skills, guided imagery, progressive relaxation, autogenic training, and the importance of physical activity to manage stress. All lessons include course assessments. During the intervention period, controls will receive weekly text messages encouraging completion of material.
  Arms: Control

SUMMARY:
The unjust social, economic, and environmental conditions that African Americans face throughout their lives lead to pervasive health disparities. These disparities are driven by healthcare differences. They are driven by economic differences. Those with less financial wealth have poorer health as compared to those with higher socioeconomic status. And yet, even when controlling for these two important social determinants of health, race still predicts morbidity and mortality.

What can account for this? Stress. African Americans experience more stress than their White peers. The story is even more dire for African American women who simultaneously face both racial discrimination and sexism. Indeed, gendered racial discrimination is nearly ubiquitous for Black women at all socioeconomic levels. It is also a distinct form of stress, with unique outcomes compared to other non-race-or-gender-related stressors. Finally, stress has clear downstream negative effects on health.

At present, there is no mobile cognitive-behavioral stress management intervention (m-CBSMi) designed to help African American women manage racial and nonracial daily stress. The investigators intend to fill this void. Using proven CBSMi techniques, participants will learn how to manage their stress through text messages and integrated mobile web content. Supportive texts will inspire, motivate, and affirm the life experiences of participants. Educational texts will increase knowledge, develop skills, and reduce barriers to adaptive coping. A library of individually tailored videos will be delivered to each participant. All mobile web content will be accessible only through touch-based links embedded within text messages, making it easy and effortless to view this material.

During Phase II the investigators will complete development of the m-CBSMi. Then, the investigators will examine the effectiveness of the m-CBSMi to reduce stress among African American female participants. Participants will be randomly assigned to either the intervention condition or to a matched control condition. Secondary measures will assess coping, well-being, subjective health, gendered racial identity, and knowledge.

ELIGIBILITY:
Inclusion Criteria:

* self-identify as Black; own a smartphone; have at least limited English literacy skills; report perceived discrimination; and be moderately stressed. The discrimination must be due to race or gender and the frequency must be at least "a few times in the past year" or more. In addition, they must report a score of 6 or higher on the 4-item Perceived Stress Scale (PSS).

Exclusion Criteria:

-

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 139 (Actual)
Dates: Start 2023-03-31 (Actual); Primary Completion 2024-05-31 (Actual); Study Completion 2024-05-31 (Actual)

PRIMARY OUTCOMES:
Change in Baseline Stress on the 10-point Perceived Stress Scale at Week 24 | Baseline and Week 24
  10-item survey that measures the degree to which an individual perceives his/her life as uncontrollable, unpredictable, and overwhelming

CONTACTS AND LOCATIONS:
Locations (1):
- ISA Associates, Alexandria, Virginia, United States

IPD SHARING:
Plan to Share IPD: Yes
The mode of dissemination of public datasets will be via archive files accessible in the public domain. Public datasets will be de-identified so that data cannot be linked to individual research participants.
Supporting Information: Study Protocol, ICF
Time Frame: Datasets will be available at a minimum once the data have been accepted for peer-reviewed publication, and earlier if the data are deemed by the PI to be clean and the sharing of data is not expected to inhibit future opportunities for publication.
Access Criteria: A data sharing agreement must be completed and signed by the requesting investigator and the Principal Investigator before this transfer of data can be made.